CLINICAL TRIAL: NCT03356834
Title: Change of Renal Function and Bone Mineral Density Marker in Chronic Hepatitis B Patients Switching From TDF to TAF vs. Maintaining TDF
Brief Title: Change of Renal Function and Bone Mineral Density in CHB Patients Switch From TDF to TAF vs. Maintaining TDF
Acronym: SWITAF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Humanity and Health Research Centre (Other)
Responsible Party: Principal Investigator, George Lau, Humanity & Healthy Medical Group President, Humanity and Health Research Centre
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HumanityHGLC
Record Dates: First submitted 2017-09-20; First posted 2017-11-29 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Chronic Hepatitis B
Keywords: Chronic hepatitis B; Efficacy, safety, and tolerability; Tenofovir alafenamide
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — tenofovir alafenamide; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TDF switch to TAF (Experimental): Tenofovir Disoproxil Fumarate(TDF) 300mg daily switch to Tenofovir Alafenamide(TAF) 25mg daily
  Interventions: Drug: Tenofovir alafenamide(TAF)
- Maintaining on TDF (Active Comparator): Maintaining on Tenofovir Disoproxil Fumarate(TDF) 300mg daily
  Interventions: Drug: Tenofovir disoproxil fumarate(TDF)

INTERVENTIONS:
Drug: Tenofovir alafenamide(TAF) — 25 mg tablet administered orally once daily
  Other Names: VEMLIDY®
  Arms: TDF switch to TAF
Drug: Tenofovir disoproxil fumarate(TDF) — 300 mg tablet administered orally once daily
  Other Names: VIREAD®
  Arms: Maintaining on TDF

SUMMARY:
In Chronic hepatitis B (CHB) patients receiving long-term sequential Neucleos(t)ides(NAs), majority of these CHB patients experienced drug resistance and switched to Tenofovir disoproxil fumaratate(TDF). However, some of patients on long term TDF experienced impairment of renal function and bone mineral density. After Tenofovir alafenamide(TAF) was in clinical practice, these group of patients got an clinical option to switch from TDF to TAF. The investigators designed a prospective cohort study to evaluate the real life effectiveness and safety in participants with chronic HBV infection switch from TDF to TAF vs. maintaining on TDF.

DETAILED DESCRIPTION:
Tenofovir disoproxil fumarate(TDF) have been associated with renal toxicity and reduced bone mineral density. Tenofovir alafenamide(TAF) is a novel tenofovir prodrug that reduces tenofovir plasma concentrations by 90%, thereby decreasing off-target side-effects. The investigators aimed to assess whether efficacy, safety, and tolerability were non-inferior in participants switched to TAF versus in those remaining on TDF. This is a prospective clinical study.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic hepatitis B,
2. Antiviral experienced,
3. Currently on long term TDF anti-HBV treatment,
4. HBV DNA < 6 log IU/ml (LLOD)
5. Able to sign the consent form of anticipating in the study

Exclusion Criteria:

1. Co-infected with HCV, HIV or other viral hepatitis,
2. Diagnosis of HCC

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 575 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Antiviral response of TAF | 60 months
  Anti-HBV effectiveness of TAF compared with TDF in treatment experienced CHB patients

SECONDARY OUTCOMES:
Improvement of renal function and bone mineral density in CHB patients switching to TAF | 60 months
  Change of renal function and bone mineral density from baseline in CHB patients of TAF a group compared with TDF group

CONTACTS AND LOCATIONS:
Locations (1):
- Humanity and Health GI and Liver Centre, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No